CLINICAL TRIAL: NCT05541003
Title: Understanding the Role of Gut Microbiota in Hyperphagia in Prader-Willi Syndrome
Acronym: PWSGUT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Keerthana Kesavarapu, D.O., Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2022000828
Record Dates: First submitted 2022-09-01; First posted 2022-09-15 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Prader-Willi Syndrome; Obesity
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm (Experimental): All participants will receive NBT-NM108 prepared as muffin (each contains 30 g of the product) for 4 weeks. The dosage will be 2 muffins a day. This dosage of NBT-NM108 will provide 24 g/day of dietary fibers.
  Interventions: Drug: NBT-NM108

INTERVENTIONS:
Drug: NBT-NM108 — All patients will consume NBT-NM108 in the form of 2 muffins daily.

SUMMARY:
This study aims to use a high-fiber supplementation, an intervention known to create shifts in the gut microbiota towards a healthier structure, to explore the relationship between gut microbiota, appetite control and feeding behavior in PWS patients.

DETAILED DESCRIPTION:
This study is recruiting PWS patients aged 18-35 years who have not received growth hormone treatment in the previous 6 months. Study candidates will be recruited from Robert Wood Johnson. Participants will attend a baseline visit at the Center for Advanced Human Brain Imaging Research (CAHBIR) at Rutgers University, during which functional magnetic resonance imaging (fMRI) coupled with a meal test will be performed to assess peripheral and central feeding pathways (7, 8). fMRI scans will be performed during resting state to assess functional connectivity of feeding related networks, with a specific focus on connectivity between the hypothalamus, insula, anterior cingulate, ventromedial/orbitofrontal prefrontal cortex and amygdala (9, 10). Activation to food (vs non-food) images will be assessed to index responsivity to appetitive feeding networks including the above regions and the ventral striatum using paradigms that have previously been found to be sensitive to trait and state in multiple studies (11-13). Thereafter participants will consume a liquid meal (525 kcal; Ensure Plus, Abbott). fMRI will be repeated immediately after the meal. Participants will obtain laboratory work coupled with a meal test to assess satiety hormones and inflammatory markers. Fasting blood draw will be taken, and the participants will consume a liquid meal (525 kcal; Ensure Plus, Abbot) followed by blood draws at 30, 60, 120, 180 and 240 min post-meal. Upon completion of baseline testing and providing a fecal sample, participants will consume NBT-NM108 (a mixture of inulin, Fibersol-2, and brans of oat, wheat, corn and sorghum; Notitia Biotechnologies) daily for 4 weeks. At the completion of the 4-week intervention, all sampling and testing will be repeated as per baseline. At baseline and end of intervention, participants will be interviewed with appetite and physical activity questionnaires (Appendix C and G) and requested to complete a 24-h food recall using MyFitnessPal, a mobile health app on their phone.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 (inclusive)
* Confirmed PWS with genetic testing
* No growth hormone treatment in the previous 6 months
* Body weight < 300 lbs.

Exclusion Criteria:

* History of other gastrointestinal disorders such as small intestinal bacterial overgrowth, celiac disease, inflammatory bowel disease, or irritable bowel syndrome.
* Pregnancy or breastfeeding
* Prior gastrointestinal or bariatric surgery
* Immunocompromised e.g., cancer treatment, bone marrow/organ transplant, immune deficiency, poorly controlled HIV/AIDS, prolonged use of steroids or other immunosuppressant medications
* Antibiotic administration in the previous 30 days
* Participation in other weight-loss programs in the previous 3 months.
* Administration of pre/probiotic supplements or antibiotics.
* Growth hormone administration in the previous 6 months
* Must have access to a smartphone, tablet, computer, or other qualifying internet-enabled device and be able to follow instructions.
* Individuals who are not proficient in English
* Contraindications for MRI scanning, including Ferrous material implanted in or on the body, including flakes or filings, surgical clips, bullets, or electrical devices such as a pacemaker, or nonremovable ferrous jewelry (fillings in teeth and permanent retainers are permitted). Individuals with surgical pins or plates above the neck are excluded. Surgical pins or plates below the neck are exclusions, except when the material is fixed to bone, and considered acceptable by the Reference Manual for Magnetic Resonance Safety. Implants and Devices, 2020 Edition. Almost all recent orthopedic implants are made of materials that are not ferromagnetic and therefore are safe for scanning, and even though some screws are still made of ferromagnetic materials these are firmly screwed into bone. In cases where the material is unknown or deemed unsafe for scanning by the Reference Manual for Magnetic Resonance Safety. Implants and Devices, the participant will be excluded. History of eye injury involving metallic materials, shavings in eyes, or welding without a face mask. Lead/iron tattoos and tattoos performed by a nonprofessional artist if the pigment material is unknown. Claustrophobia (history of significant anxiety in closed places).
* Back problem that would prevent the subject from laying still comfortably for up to 60 minutes.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holland AJ, Treasure J, Coskeran P, Dallow J, Milton N, Hillhouse E. Measurement of excessive appetite and metabolic changes in Prader-Willi syndrome. Int J Obes Relat Metab Disord. 1993 Sep;17(9):527-32. PMID 8220655
- [Background] Fieldstone A, Zipf WB, Sarter MF, Berntson GG. Food intake in Prader-Willi syndrome and controls with obesity after administration of a benzodiazepine receptor agonist. Obes Res. 1998 Jan;6(1):29-33. doi: 10.1002/j.1550-8528.1998.tb00311.x. PMID 9526967
- [Background] Proffitt J, Osann K, McManus B, Kimonis VE, Heinemann J, Butler MG, Stevenson DA, Gold JA. Contributing factors of mortality in Prader-Willi syndrome. Am J Med Genet A. 2019 Feb;179(2):196-205. doi: 10.1002/ajmg.a.60688. Epub 2018 Dec 19. PMID 30569567
- [Background] Martinez Michel L, Haqq AM, Wismer WV. A review of chemosensory perceptions, food preferences and food-related behaviours in subjects with Prader-Willi Syndrome. Appetite. 2016 Apr 1;99:17-24. doi: 10.1016/j.appet.2015.12.021. Epub 2015 Dec 20. PMID 26713776
- [Background] Zhang C, Yin A, Li H, Wang R, Wu G, Shen J, Zhang M, Wang L, Hou Y, Ouyang H, Zhang Y, Zheng Y, Wang J, Lv X, Wang Y, Zhang F, Zeng B, Li W, Yan F, Zhao Y, Pang X, Zhang X, Fu H, Chen F, Zhao N, Hamaker BR, Bridgewater LC, Weinkove D, Clement K, Dore J, Holmes E, Xiao H, Zhao G, Yang S, Bork P, Nicholson JK, Wei H, Tang H, Zhang X, Zhao L. Dietary Modulation of Gut Microbiota Contributes to Alleviation of Both Genetic and Simple Obesity in Children. EBioMedicine. 2015 Jul 10;2(8):968-84. doi: 10.1016/j.ebiom.2015.07.007. eCollection 2015 Aug. PMID 26425705
- [Background] Purtell L, Sze L, Loughnan G, Smith E, Herzog H, Sainsbury A, Steinbeck K, Campbell LV, Viardot A. In adults with Prader-Willi syndrome, elevated ghrelin levels are more consistent with hyperphagia than high PYY and GLP-1 levels. Neuropeptides. 2011 Aug;45(4):301-7. doi: 10.1016/j.npep.2011.06.001. Epub 2011 Jul 1. PMID 21722955
- [Background] Dykens EM, Maxwell MA, Pantino E, Kossler R, Roof E. Assessment of hyperphagia in Prader-Willi syndrome. Obesity (Silver Spring). 2007 Jul;15(7):1816-26. doi: 10.1038/oby.2007.216. PMID 17636101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment time period was from 11/1/2022 to 3/1/2023. Recruitment occurred from Robert Wood Johnson medical clinics.
Pre-assignment Details: No patients were excluded from the study before assignment to arms or groups.
Period: Overall Study
Arm/Group | Experimental Arm
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Fiber Intervention: All patients were given 48 grams of NBT-NM108 dietary fiber in the form of 2 muffins per day
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Weight [Mean (Standard Deviation); unit: kilogram] — Weight of individual before fiber intervention.
  kilogram | 107.01 (21.33)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 38.58 (7.82)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 135 (13.64)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 88.91 (9.63)
Heart Rate [Mean (Standard Deviation); unit: Beats per minute] | 81.55 (15.92)

OUTCOME MEASURES:

1. Primary Outcome: Microbiome Analysis: Alpha Diversity
Description: Alpha Diversity measured by Shannon index. The Shannon Index is a measure of diversity of microbial species that takes into account both abundance (the number of species present) and evenness (how close the numbers for each species are). The Shannon index can be calculated using the following equation: H= -∑(i=1)^s pi ln(pi). A value of zero for H indicates that a community has only one species. The higher the value of H, the higher the diversity of species in a particular community.
Time Frame: Weeks 0
Population: Alpha Diversity measured by Shannon index. The Shannon Index is a measure of diversity of microbial species that takes into account both abundance (the number of species present) and evenness (how close the numbers for each species are). The Shannon index can be calculated using the following equation: H= -∑(i=1)^s pi ln(pi). A value of zero for H indicates that a community has only one species. The higher the value of H, the higher the diversity of species in a particular community. No units.
Measure: Mean (Standard Deviation); unit: Shannon index
Groups:
- Microbiome Structure: In this pilot study, we collected 20 fecal samples from 10 subjects before and after the dietary intervention. We extracted the metagenomic DNA from the fecal samples and applied 16S rRNA gene amplicon sequencing to understand the impact of NBT-NM108 on the gut microbiome. We obtained ~980,000 high-quality sequencing reads from 20 samples and have identified 757 amplicon sequence variants (ASVs) from these samples. For subsequent analysis the number of sequencing reads per sample was normalized to 34,000 per sample. Alpha and beta diversity were analyzed to assess changes of the overall gut microbiota structure. Alpha diversity describes the overall gut microbiota structure within a single sample.
Arm/Group | Microbiome Structure
Number analyzed (Participants) | 10
Shannon index | 4.89 (0.46)

2. Primary Outcome: Microbiome Analysis: Alpha Diversity
Description: Alpha diversity measured by Shannon index. "The Shannon Index is a measure of diversity of microbial species that takes into account both abundance (the number of species present) and evenness (how close the numbers for each species are). The Shannon index can be calculated using the following equation: H= -∑(i=1)^s pi ln(pi). A value of zero for H indicates that a community has only one species. The higher the value of H, the higher the diversity of species in a particular community.
Time Frame: Week 4
Population: For alpha diversity, Shannon index was used.
Measure: Mean (Standard Deviation); unit: Shannon index
Groups:
- Microbiome Structure: Alpha Diversity: For alpha diversity, Shannon index and observed number of ASVs were used for assessment. Both the indices were computed for each sample and are represented as Mean (Standard deviation).
Arm/Group | Microbiome Structure: Alpha Diversity
Number analyzed (Participants) | 10
Shannon index | 4.73 (0.41)

3. Primary Outcome: Microbiome Analysis: Beta Diversity
Description: The Bray-Curtis distance was used to compute the distances for each sample. Bray-Curtis distance uses species abundance information and membership to calculate the distance between samples. The Bray-Curtis dissimilarity index for a sample ranges between 0 and 1. A value of 0 indicates no difference between the samples, while a value of 1 represents the maximum distance between them
Time Frame: Week 0
Population: For beta diversity, Bray-Curtis dissimilarity index was computed for each sample. Bray-Curtis dissimilarity index is represented as Median (Inter-Quartile Range).
Measure: Median (Inter-Quartile Range); unit: Bray-Curtis distance
Groups:
- Microbiome: Beta Diversity: For beta diversity, Bray-Curtis dissimilarity index was computed for each sample. Bray-Curtis dissimilarity index is represented as Median (Inter-Quartile Range).
Arm/Group | Microbiome: Beta Diversity
Number analyzed (Participants) | 10
Bray-Curtis distance | 0.76 [0.65 to 0.81]

4. Secondary Outcome: Weight
Description: Weight in kg
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
Kilogram | 107 (22)

5. Secondary Outcome: Acyl-Ghrelin Level
Description: Early response to meal post-intervention is 0-30min. Late response phase to meal post-intervention is 60-180min.
Time Frame: Week 0
Population: Looking at iAUC for early and late response phases after meal.
Measure: Mean (Standard Deviation); unit: pg*min/mL
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
pg*min/mL
  Early Response | 13.47 (22.54)
  Late Response | 187 (191)

6. Secondary Outcome: Acyl-Ghrelin Level
Description: Early response to meal post-intervention is 0-30min. Late response phase to meal post-intervention is 60-180min.
Time Frame: Week 4
Population: Looking at iAUC for early and late response phases after meal.
Measure: Mean (Standard Deviation); unit: pg*min/mL
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
pg*min/mL
  Early Response | 12.5 (17.6)
  Late Response | 278 (605)

7. Secondary Outcome: Peptide YY (PYY)
Description: Early response to meal post-intervention is 0-30min. Late response phase to meal post-intervention is 60-180min.
Time Frame: Week 0
Population: Looking at iAUC for early and late response phases after meal.
Measure: Mean (Standard Deviation); unit: pg*min/mL
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
pg*min/mL
  early phase (0-30min) | 0.23 (0.37)
  late phase response (60-180min) | 4.01 (4.22)

8. Secondary Outcome: Peptide YY (PYY)
Description: Early response to meal post-intervention is 0-30min. Late response phase to meal post-intervention is 60-180min.
Time Frame: Week 4
Population: Looking at iAUC for early and late response phase after meal.
Measure: Mean (Standard Deviation); unit: pg*min/mL
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
pg*min/mL
  early phase (0-30min) | 0.614 (1.43)
  late phase response (60-180min) | 11.1 (14.1)

9. Secondary Outcome: Glucagon Like Peptide 1 (GLP1)
Description: GLP1 levels were measured in patients before fiber intervention. Early response to meal post-intervention is 0-30min. Late response phase to meal post-intervention is 60-180min.
Time Frame: Week 0
Population: Looking at iAUC for early and late response phase after meal.
Measure: Mean (Standard Deviation); unit: pg*min/ml
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
pg*min/ml
  early phase (0-30min) | 10.6 (15.8)
  late phase response (60-180min) | 115 (184)

10. Secondary Outcome: Glucagon Like Peptide 1 (GLP1)
Description: GLP1 levels were measured in patients after fiber intervention. Early response to meal post-intervention is 0-30min. Late response phase to meal post-intervention is 60-180min.
Time Frame: Week 4
Population: Looking at iAUC for early and late response phase after meal.
Measure: Mean (Standard Deviation); unit: pg*min/ml
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
pg*min/ml
  early phase (0-30min) | 4.44 (6.85)
  late phase response (60-180min) | 79.6 (55.7)

11. Secondary Outcome: Insulin Level
Description: Insulin levels were measured in patients before fiber intervention. Early response to meal post-intervention is 0-30min. Late response phase to meal post-intervention is 60-180min.
Time Frame: Week 0
Population: Looking at iAUC for early and late response phase after meal.
Measure: Mean (Standard Deviation); unit: µIU*min/ml
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
µIU*min/ml
  early phase (0-30min) | 1660 (716)
  late phase response (60-180min) | 6361 (3978)

12. Secondary Outcome: Insulin Level
Description: Insulin levels were measured in patients after fiber intervention. Early response to meal post-intervention is 0-30min. Late response phase to meal post-intervention is 60-180min.
Time Frame: Week 4
Population: Looking at iAUC for early and late response phase after meal.
Measure: Mean (Standard Deviation); unit: µIU*min/ml
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
µIU*min/ml
  early phase (0-30min) | 1607 (783)
  late phase response (60-180min) | 7427 (3644)

13. Secondary Outcome: Glucose Level
Description: Glucose levels were measured in patients before fiber intervention. Early phase (0-30min) and late phase response (60-180min) to a mixed meal tolerance test was collected.
Time Frame: Week 0
Population: Looking at iAUC for early and late response phase after meal.
Measure: Mean (Standard Deviation); unit: mmol*min/mL
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
mmol*min/mL
  early phase (0-30min) | 264 (288)
  late phase response (60-180min) | 301 (503)

14. Secondary Outcome: Glucose Level
Description: Glucose levels were measured in patients after fiber intervention. Early phase (0-30min) and late phase response (60-180min) to a mixed meal tolerance test was collected.
Time Frame: Week 4
Population: Glucose levels were measured in patients after fiber intervention. Early phase (0-30min) and late phase response (60-180min) to a mixed meal tolerance test was collected.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
mmol/L
  early phase (0-30min) | 182 (222)
  late phase response (60-180min) | 375 (552)

15. Secondary Outcome: Calorie Count
Description: 24 hour dietary recall recorded in MyFitnessPal application measured in kcal.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: Kcal
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 12
Kcal | 1638 (493)

16. Secondary Outcome: Calorie Count
Description: 24 hour dietary recall recorded in MyFitnessPal application measured in kcal.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Kcal
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
Kcal | 1840 (564)

17. Secondary Outcome: Hyperphagia Questionnaire
Description: Appetite behavior measured by questionnaire measured by likert scale. The scores should improve from week 0 to week 4. Higher scores indicate worse hyperphagia.
Time Frame: Week 0
Population: The questionnaire includes 11 questions measured on a 5-point Likert scale, which are summarized in a total hyperphagia score (range: 11-55). Three subscores were summed: hyperphagic behavior (range: 5-25), hyperphagic drive (range: 4-20) and hyperphagic severity (range: 2-10). The scores should improve from week 0 to week 4 with intervention. Higher scores indicate worse hyperphagia. Our scores reported below are mean +/- standard deviation and not ranges.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 12
scores on a scale
  Hyperphagia behavior | 6.18 (1.83)
  Hyperphagia drive | 6.54 (2.20)
  Hyperphagia severity | 3.63 (1.69)

18. Secondary Outcome: Hyperphagia Questionnaire
Description: Appetite behavior measured by questionnaire measured by likert scale. The scores should improve from week 0 to week 4. Higher scores indicate worse hyperphagia. The questionnaire includes 11 questions measured on a 5-point Likert scale, which are summarized in a total hyperphagia score (range: 11-55). Three subscores were summed: hyperphagic behavior (range: 5-25), hyperphagic drive (range: 4-20) and hyperphagic severity (range: 2-10). The scores should improve from week 0 to week 4 with intervention. Higher scores indicate worse hyperphagia.
Time Frame: Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fiber Intervention
Number analyzed (Participants) | 10
scores on a scale
  Hyperphagia behavior | 5.3 (1.7)
  Hyperphagia drive | 5.7 (1.7)
  Hyperphagia severity | 3.1 (1.4)

19. Primary Outcome: Microbiome Analysis: Beta Diversity
Description: as for outcome 3
Time Frame: Week 4
Population: For beta diversity, Bray-Curtis dissimilarity index was computed for each sample.
Measure: Median (Inter-Quartile Range); unit: Bray-Curtis distance
Arm/Group | Microbiome: Beta Diversity
Number analyzed (Participants) | 10
Bray-Curtis distance | 0.73 [0.64 to 0.79]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Patients are asked to keep a supplement log. On this log patients record if and when they take the fiber supplement and any side effects. Only 10 participants took fiber supplement.
Arm/Group | Fiber Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
There was a variance in BMI in patients accepted. We anticipate this led the varied difference in response in data. Additionally, two of the patients had PWS while the remainder of patients had non-genetic obesity. We anticipate this also led to the varied difference in response in data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT05541003/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT05541003/ICF_002.pdf